CLINICAL TRIAL: NCT04880070
Title: Post Market Clinical Follow Up Study to Collect Additional Data and Imaging
Brief Title: Post-Market Clinical Follow Up Study to Collect Additional Data and Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SW-MCPM-2021
Record Dates: First submitted 2021-05-05; First posted 2021-05-10 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Connective Tissue Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Shockwave Device (Experimental): The Shockwave device will be used on multiple areas of the body for the purpose of treating connective tissue.
  Interventions: Device: Shockwave Treatment

INTERVENTIONS:
Device: Shockwave Treatment — Self-controlled, single-arm group using the Shockwave device.

SUMMARY:
This is a prospective, open label, multi-center clinical study to collect additional data and imaging for the ViaSure device.The intended use of the ViaSure device used in this study is to assess the usability and tissue response to shock wave treatment.

DETAILED DESCRIPTION:
Up to 50 subjects will be enrolled at 2 study centers. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 5 treatments with the study device. Follow up visits may occur 30 and 90 days post last treatment visit.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female 18 - 65 years of age.
* Willing to undergo treatments with the SoftWave device.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject has a pacemaker or implantable defibrillator.
* The subject has a severe coagulation disorder.
* The subject has open epiphyseal plates.
* The subject has recently had a steroid injection.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months to entering this study.
* The subject has any condition or is in a situation which, in the Investigator's opinion, may put the subject at significant risk, may

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2021-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (1):
- Cynosure, Inc., Westford, Massachusetts, United States

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Shockwave Device
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Shockwave Device
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 5
FitzPatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Types range from I-VI, with I being low melanin content (lighter skin), and VI being high melanin content (darker skin). The reference provided in the references section gives more details if needed.
  Participants
    Fitzpatrick Skin Type I | 1
    Fitzpatrick Skin Type II | 2
    Fitzpatrick Skin Type III | 2
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 0

OUTCOME MEASURES:

1. Primary Outcome: # of Subjects With Altered Gene Expression
Description: Subjects had their gene expression relative to their own baseline samples analyzed using nSolver 4.0 software, and this was done 14 days post treatment.
Time Frame: 14 days post treatment
Population: 1 subject did not have their 14 day sample analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Shockwave Device
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: Subjects had their adverse events tracked from the beginning of the study to 14 days post treatment.
Arm/Group | Shockwave Device
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT04880070/Prot_SAP_000.pdf